CLINICAL TRIAL: NCT05630573
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase Ib/IIa Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of TNM001 Injection in Chinese Healthy Preterm and Term Infants
Brief Title: A Study of TNM001 in Chinese Healthy Preterm and Term Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNM001-201
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TNM001 Injection dose 1 (Experimental): low dose administered
  Interventions: Biological: TNM001
- TNM001 Injection dose 2 (Experimental): medium dose administered
  Interventions: Biological: TNM001
- TNM001 Injection dose 3 (Experimental): high dose administered
  Interventions: Biological: TNM001
- placebo (Placebo Comparator): placebo administered
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TNM001 — intramuscular injection
  Arms: TNM001 Injection dose 1; TNM001 Injection dose 2; TNM001 Injection dose 3
Biological: Placebo — intramuscular injection
  Arms: placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability and pharmacokinetics (PK) profile of TNM001 injection in healthy preterm and term infants. The main questions it aims to answer are:

* the safety and tolerability of TNM001 injection
* the pharmacokinetic (PK) profile of TNM001

DETAILED DESCRIPTION:
This phase Ib/IIa study is designed to assess the safety, tolerability, and pharmacokinetics (PK) profile TNM001 in healthy preterm and term infants. This study will also compare the incidence of Respiratory Syncytial Virus（RSV） infection between different doses of TNM001 and placebo, which will be used to select the dose to be studied in the later phase of clinical trials of TNM001. Approximately 30 subjects will be randomized and will be dosed once on Day 1 and followed up until Day 151. Around 6 investigational study centres participate in the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy preterm infants and term infants within 1 year old of age
2. Infants who are in the first RSV infection season at the time of randomization

Key Exclusion Criteria:

1. Any fever or acute illness within 7 days prior to dosing
2. LRTI prior to randomization
3. Received any anti-RSV monoclonal antibody or RSV vaccine
4. Any other circumstances that, in the opinion of the investigator, may interfere with the assessment of the study drug or the interpretation of the study results
5. The subject is a child of the investigator or his/her subordinate study personnel or relatives or sponsor staff

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TNM001 Injection | 150 days post dose
  Type and incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) of TNM001 | 150 days post dose
  The pharmacokinetic (PK) parameter AUC (0-infinity) will be estimated based on the serum concentrations of TNM001
Maximum Observed Serum Concentration (Cmax) of TNM001 | 150 days post dose
  The Cmax is the maximum observed serum concentration of TNM001
Terminal Elimination Half Life (t1/2) of TNM001 | 150 days post dose
  Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the serum
Serum anti-RSV neutralizing antibodies titer levels in each dose cohort | 150 days post dose
  To summarize the proportion of subjects with severalfold increase after dosing compared to the predose (baseline)
Anti-drug antibody (ADA) positive rate of TNM001 | 150 days post dose
  The evaluation indicator of immunogenicity is the ADA positive rate in subjects

OTHER OUTCOMES:
Lower respiratory tract infection(LRTI) | 150 days post dose
  The incidence of LRTI

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Liu, Principal Investigator — West China Second Hospital, Sichuan University; Qin Yu, Principal Investigator — West China Second Hospital, Sichuan University
Locations (6):
- China (6):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Linfen People's Hospital, Linfen, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided